CLINICAL TRIAL: NCT00170014
Title: Reproducibility of Magnetocardiography Measurements Using the Cardiomag Magnetocardiograph System Model 2409 and Its Software for Data Acquisition and Analysis
Brief Title: Precision of the Magnetocardiographer for Data Aquision and Analysis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: CardioMag Imaging (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 850-04
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

INTERVENTIONS:
Device: Magnetocardiograph

SUMMARY:
magnetocardiography has been extensively studied focusing on the possible clinical applications of the device. Evaluating the precision of a device is a prerequisite condition to know what are significant changes and how can these be trusted. A respectable reproducibility study for the MCG measurements is crucial for this new device to be used for clinical applications. In this study, we will focus on a critical portion of the heart cycle assessing for changes in time of the computerized analysis of this phase and comparing the analysis done by two examiners.

DETAILED DESCRIPTION:
The studies involving magnetocardiography have almost exclusively focused on evaluating possible clinical applications of the device. Leder et al saw the need for investigating the reproducibility of High Temperature Superconducting (HTS-)MCG measurements. They tested 18 healthy volunteers, stating that assessment of the reproducibility of HTS-MCGs in the normal heart is a prerequisite condition for the definition of significant levels of changes which, for instance, may be observed in serial measurements of patients suffering from acute coronary syndromes. They also pointed out the potentially strong electromagnetic interference inside a hospital, likely to be very different from the noise found in engineering laboratories where the MCGs are originally calibrated and tested. A respectable reproducibility for the MCG measurements is crucial for clinical applications. Leder et al studied the reproducibility of QRS complexes, ST segments, and T waves. They found that the reproducibility of the measurements in the depolarization phase was high, whereas the reproducibility of their repolarization readings was considerably lower. The results led Leder et al to conclude that further technical development was needed to improve signal-to-noise ratio allowing for clinical application of repolarization abnormalities for recognizing Acute Coronary Syndromes. In this study, we will focus on the repolarization phase by assessing the reproducibility of the T wave only. Comparison of scores and results based on computer analyses will provide the basis for our evaluation. Visual interpretations by the two examiners will also be compared.

ELIGIBILITY:
Age less than or equal to 45 years

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The objective of our study is to evaluate inter-examiner reproducibility in the MCG results retrieved from data acquisition and analysis by two examiners. HTS-MCG measurements will be obtained from healthy AND diseased subjects in an unshielded clinical

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Smars, M.D. EM, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States